CLINICAL TRIAL: NCT06338137
Title: Comparison of High and Low Pulse Energy Dusting Protocols Using Holmium: YAG-laser in Flexible Ureteroscopy for Renal Stones Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Hossam Kandeel, Director, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2024urol
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis | interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-energy patients (Other): Use high energy in stone management
  Interventions: Device: Holmium Yag laser
- Low energy patient (Other): Use low energy in stone management
  Interventions: Device: Holmium Yag laser

INTERVENTIONS:
Device: Holmium Yag laser — Use two laser energy low and high to reach the optimal setting for stone dusting

SUMMARY:
Rcompare high-energy versus low-energy laser settings in renal stone lithotripsy using low power machines) Holmium YAG 30 watts, examining their respective advantages, limitations, and overall efficacy.

DETAILED DESCRIPTION:
The prevalence of urinary stone disease treatment has shown a continuous updating Within the armamentarium of urinary stone management, the laser has emerged as a cornerstone for lithotripsy in endourological procedures. The laser technology has witnessed a progressive evolution, transitioning from the established holmium: yttrium-aluminum-garnet (Ho:YAG) laser with pulse modulation to the advent of thulium fiber laser (TFL) and, more recently, the innovative pulsed thulium:YAG (p-Tm:YAG) laser Laser lithotripsy is prefered for its minimally invasive approach and high success rates in fragmenting stones, yet the ongoing debate continues regarding the optimal laser power settings for this procedure. contemporary approaches in laser lithotripsy focus on two primary strategies: fragmenting stones into smaller retrievable parts or breaking them into minute fragments, commonly referred to as 'dust,' facilitating the natural passage of smaller particles The choice between high power and low power settings in laser lithotripsy significantly influences treatment outcomes, including stone fragmentation efficiency, procedural time, and potential tissue damage. High-energy power laser settings offer rapid stone ablation capabilities, enabling quick fragmentation but potentially raising concerns about thermal injury to surrounding tissues. In contrast, low-energy power settings, while reducing the risk of tissue damage, might prolong the procedure and necessitate additional maneuvers for complete stone clearance This study aims to compare high-energy versus low-energy laser settings in renal stone lithotripsy using low power machines) Holmium YAG 30 watts, examining their respective advantages, limitations, and overall efficacy. By scrutinizing existing literature and recent studies, this study intends to provide a 56 comprehensive understanding of the clinical implications of choosing optimal laser settings in urolithiasis comprehensive understanding of the clinical implications of choosing optimal laser settings in urolithiasis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* hard renal stones
* less than 2 cm
* Hounsfield unit of ≥ 1000

Exclusion Criteria:

* Patients less than 18 years
* ureteral stones
* stones with Hounsfield units less than 1000
* stones in calyceal diverticulum
* patients with coagulopathy were also excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Stone free rates | One year
  Assess stone free rate between two different setting

SECONDARY OUTCOMES:
Preoperative complications | One year
  To assess complications between low and high energy

CONTACTS AND LOCATIONS:
Locations (1):
- Hossam Kandeel, Shibīn al Kawm, State Or Province, Egypt